CLINICAL TRIAL: NCT06888622
Title: Eculizumab for Blaze-limiting Approach in NMOSD: A Prospective Study
Brief Title: BLAZE-Limiting Approach in NMOSD
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chao Quan, Professor, Chief Physician, Huashan Hospital
Other Study IDs: KY2025-062; MR-31-22-008563; ChiCTR2000030 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorders (NMOSD)
Keywords: NMOSD; eculizumab; AQP4-ab; Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eculizumab treatment group: Eculizumab was administered intravenously at a dosage of 900 mg weekly for four consecutive weeks
  Interventions: Drug: Eculizumab administration

INTERVENTIONS:
Drug: Eculizumab administration — Eculizumab was administered intravenously at a dosage of 900 mg weekly for four consecutive weeks

SUMMARY:
This is an observational cohort study based on data from the hospital-based NMOSD registry (Chinese Medical Research Registration Number MR-31-22-008563; ChiCTR2000030651). Between October 2023 (when eculizumab was approved for NMOSD in China) and February 2025, 26 consecutive patients with AQP4-IgG-positive NMOSD received eculizumab, and 9 of them were included in this study.

ELIGIBILITY:
Inclusion Criteria:

(1)Patients have been diagnosed with NMOSD and tested seropositive for AQP4 antibody; (2) Age ≥ 18 years; (3) Received eculizumab during an acute phase of NMOSD, defined as within 30 days of attack onset； (4) Adherence to an 8-week follow-up from eculizumab initiation.

Exclusion Criteria:

1. Patients with unresolved Neisseria meningitidis infection or severe infections that preclude the use of immunotherapy;
2. Patients with severe comorbidities (such as heart failure, respiratory failure, severe hepatic or renal dysfunction, etc.);
3. Patients with incomplete records of clinical symptoms and signs, as well as insufficient data on serum marker tests in their medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational cohort study based on data from the prospectively followed NMOSD cohort of the hospital-based registry (The Chinese Medical Research Registration Number MR-31-22-008563; ChiCTR2000030651). Between October 2023 (when eculizumab was approved for NMOSD in China) and February 2025 consecutive patients with AQP4-IgG-positive NMOSD received eculizumab were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
The change in disability status measured by the MRC scale score | 0, 1, 2, 3, 4, 8 weeks
  Measured by the MRC scale score for patients with LETM
The change in disability status | 0, 1, 2, 3, 4, 8 weeks
  Measured by the best corrected visual acuity (BCVA)

SECONDARY OUTCOMES:
Incidence of AEs and SAEs during eculizumab treatment | 1, 2, 3, 4, 8 weeks
  dverse events were coded using MedDRA version 27.1. Adverse events were analyzed in the safety analysis population (all patients who received at least one dose of study treatment) in terms of percentage incidence and as rates by exposure time (number of events per 100 patient-years of exposure and the associated 95% CI) to adjust for any differences in duration of exposure. The severity of adverse events was measured by NCI CTCAE version 5.0.
The Change in Expanded Disability Status Scale (EDSS) scores | 0, 1, 2, 3, 4, 8 weeks
  Measured by Expanded Disability Status Scale (EDSS) scores for the entire cohort.
The Change in Opticospinal Impairment Scale (OSIS) scores | 0, 1, 2, 3, 4, 8 weeks
  Measured by Opticospinal Impairment Scale (OSIS) for the entire cohort.
The change in Visual Functional System Score (VFSS) | 0, 1, 2, 3, 4, 8 weeks
  Measured by Visual Functional System Score (VFSS) for patients with ON.

OTHER OUTCOMES:
The changes of serological biomarkers (sGFAP and sNfL) | 0, 2, 4, 8 weeks
  Serum GFAP and NfL concentrations were analyzed in duplicates using SIMOA.
The changes of OCT measurements (pRNFL and mGCIPL). | 0, 1, 2, 3, 4, 8 weeks
  The peripapillary retinal nerve fiber layer (pRNFL) and macular ganglion cell-inner plexiform layer (mGCIPL) was analyzed by optical coherence tomography (OCT) measurements

CONTACTS AND LOCATIONS:
Overall Officials: Chao Quan, Doctor, Principal Investigator — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No